CLINICAL TRIAL: NCT01893515
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled 12-Week Phase II Proof of Concept Study to Evaluate the Efficacy and Safety of PRC-4016 Once Daily Versus Placebo in Statin-Naïve or Statin-Stable Hypertriglyceridemic Subjects
Brief Title: The Efficacy and Safety of PRC-4016 in Hypertriglyceridemic Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pronova BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTN 4016 13201
Record Dates: First submitted 2013-06-28; First posted 2013-07-09 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PRC-4016 (Experimental): PRC-4016, oral administration once daily, capsule
  Interventions: Drug: PRC-4016
- Placebo (Placebo Comparator): Placebo, oral administration once daily, capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRC-4016
  Arms: PRC-4016
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objectives of this study is

* To evaluate the efficacy of PRC-4016 by assessment of the percentage change in blood lipids and lipoprotein parameters from baseline after 12 weeks of treatment.
* To evaluate the safety of PRC-4016 as assessed by adverse events and other safety parameters

DETAILED DESCRIPTION:
6-8 weeks screening period with diet/lifestyle stabilization and lipid qualification

ELIGIBILITY:
Main Inclusion Criteria:

* Fasting triglycerides 500-1500 mg/dl
* Not on other lipid altering therapy, OR on stable lipid altering therapy

Main Exclusion Criteria:

* Type I diabetes or uncontrolled type II diabetes
* Recent cardiovascular or coronary event
* History of pancreatitis
* History or evidence of major and clinically significant diseases that would interfere with the conduct of the study or interpretation of data
* Uncontrolled hypertension

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Percent change in triglycerides from baseline to week 12 | from baseline to Week 12

SECONDARY OUTCOMES:
Change in HDL-C from baseline to Week 12 | from baseline to Week 12
Change in non-HDL-C from baseline to Week 12 | from baseline to Week 12
Change in LDL-C from baseline to Week 12 | from baseline to week 12
Change in VLDL-C from baseline to Week 12 | from baseline to week 12
Change in total cholesterol from baseline to Week 12 | from baseline to week 12
Change in ApoA1 from baseline to Week 12 | from baseline to Week 12
Change in Apo B from baseline to Week 12 | from baseline to week 12
Change in insulin from baseline to Week 12 | from baseline to Week 12
Change in fasting plasma glucose from baseline to Week 12 | from baseline to Week 12
Change in HbA1c from baseline to Week 12 | from baseline to Week 12
Change in insulin resistance (HOMA) from baseline to Week 12 | from baseline to Week 12
Change in Lp-PLA2 from baseline to Week 12 | from baseline to Week 12
Change in hsCRP from baseline to Week 12 | from baseline to Week 12
Change in red blood cell content of EPA and DHA from baseline to Week 12; | from baseline to Week 12;

OTHER OUTCOMES:
Safety assessments will include adverse events, clinical laboratory measurements (chemistry, hematology, and urinalysis), 12-lead ECGs, blood pressure, and physical examinations. | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pål Nord, MD, MPH, Study Director — Pronova BioPharma; Traci A. Turner, MD, MT, Principal Investigator — Metabolic and Atherosclerosis Research Center
Locations (39):
- United States (39):
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Terence Hart, MD, Muscle Shoals, Alabama
  - Central Phoenix Medical Clinic, Phoenix, Arizona
  - Pacific Oaks Medical Group, Beverly Hills, California
  - National Research Institute - Wilshire, Los Angeles, California
  - National Research Institute - East 118, Los Angeles, California
  - Research Across America - Santa Ana, Santa Ana, California
  - Encompass Clinical Research, Spring Valley, California
  - Colorado Springs Health Partners, Colorado Springs, Colorado
  - Clinical Research of South Florida, Coral Gables, Florida
  - Jacksonville Impotence Treatment Center, Jacksonville, Florida
  - Compass Research East, LLC, Oviedo, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Meridien Research, St. Petersburg, Florida
  - Meridien Research- Tampa, Tampa, Florida
  - Evanston Premier Healthcare Research LLC, Evanston, Illinois
  - Medisphere Medical Research Center, Evansville, Indiana
  - Heartland Research Assoc., LLC, Newton, Kansas
  - Louisville Metabolic and Atherosclerosis Research Center (L-MARC), Louisville, Kentucky
  - Troy Internal Medicine, P.C., Troy, Michigan
  - Radiant Research - Edina, Edina, Minnesota
  - Mercury Street Medical, Butte, Montana
  - Peters Medical Research, High Point, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - PMG Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Sterling Research Group, Ltd. - Auburn, Cincinnati, Ohio
  - Metabolic and Atherosclerosis Research Center, Cincinnati, Ohio
  - Columbus Clinical Research, Inc., Columbus, Ohio
  - PSB Research/P. S. Bains, M.S., D.O., Marion, Ohio
  - RAS Health Ltd, Marion, Ohio
  - Lynn Health Science Institute - Oklahoma City, Oklahoma City, Oklahoma
  - Willamette Valley Clinical Studies, Eugene, Oregon
  - Green and Seidner Family Practice Associates, Lansdale, Pennsylvania
  - UnitedResearch - Orangeburg, LLC, Orangeburg, South Carolina
  - Padre Coast Clinical Research, Corpus Christi, Texas
  - Advanced Clinical Research, West Jordan, Utah
  - National Clinical Research - Norfolk, Inc., Norfolk, Virginia
  - National Clinical Research - Richmond, Inc., Richmond, Virginia

REFERENCES:
- [Derived] Bays HE, Hallen J, Vige R, Fraser D, Zhou R, Hustvedt SO, Orloff DG, Kastelein JJ. Icosabutate for the treatment of very high triglycerides: A placebo-controlled, randomized, double-blind, 12-week clinical trial. J Clin Lipidol. 2016 Jan-Feb;10(1):181-91.e1-2. doi: 10.1016/j.jacl.2015.10.012. Epub 2015 Nov 14. PMID 26892135